CLINICAL TRIAL: NCT06076850
Title: Extracorporeal Shockwave Therapy for Penile Rehabilitation in Post-Radical Prostatectomy Patients: A Randomized, Double-Blinded, Sham-Controlled Study
Brief Title: Low-Intensity Extracorporeal Shockwave Therapy for Penile Rehabilitation in Post-Radical Prostatectomy Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Pengajar Universiti Putra Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JKEUPM-2023-073
Record Dates: First submitted 2023-07-23; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Erectile Dysfunction Following Radical Prostatectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care + Active LiESWT (Active Comparator): Tadalafil 5mg daily - to start 5 days before surgery and continued for 12 months after surgery till end of study.
  With or without Vacuum Pump
  Active LiESWT
  Interventions: Device: Low-Intensity Extracorporeal Shockwave Therapy (LiEWST) - Active
- Standard Care + Sham LiESWT (Sham Comparator): Tadalafil 5mg daily - to start 5 days before surgery and continued for 12 months after surgery till end of study.
  With or without Vacuum Pump
  Sham LiESWT
  Interventions: Device: Low-Intensity Extracorporeal Shockwave Therapy (LiEWST) - Sham

INTERVENTIONS:
Device: Low-Intensity Extracorporeal Shockwave Therapy (LiEWST) - Active — Treatment protocol:
  * EFD 0.096 mJ/mm2
  * 2 sessions / week; 5000 shocks / session
  * 6 weeks treatment
  * total: 12 sessions
  * Li-ESWT to start after removal of indwelling catheter
  Other Names: Dornier Aries 2 (Dornier MedTech, Germany)
  Arms: Standard Care + Active LiESWT
Device: Low-Intensity Extracorporeal Shockwave Therapy (LiEWST) - Sham — Treatment protocol:
  * EFD 0 mJ/mm2
  * 2 sessions / week; 5000 shocks / session
  * 6 weeks treatment
  * total: 12 sessions
  * Li-ESWT to start after removal of indwelling catheter
  Other Names: Dornier Aries 2 (Dornier MedTech, Germany)
  Arms: Standard Care + Sham LiESWT

SUMMARY:
Radical prostatectomy (RP) is one of the curative treatment modalities for localized or locally advanced prostate cancer. Urinary incontinence and erectile dysfunction (ED) are two most common complications after RP. Despite the advancement of prostate cancer treatment, ED post-RP remains a significant morbidity especially for patients who are sexually active pre-operatively. To improve the sexual function post-surgery, numerous strategies have been described including preservation of neurovascular bundles intra-operatively, post-operative physiotherapy, on-demand phosphodiesterase 5-inhibitors (PDE5i), regular PDE5i, intra-carvenosal injection or vacuum suction device.

Low-intensity extracorporeal shockwave therapy (LiESWT) is an emerging treatment modality of ED with promising result, and it is a well-established treatment of ED in patients with diabetes mellitus or vasculopathy. Most of the pre-clinical studies were done on post-RP ED rat models with bilateral cavernous nerve crush injury. LiESWT was observed to improve nerve-impaired ED significantly compared to sham procedures. There are currently one pilot study and one randomized controlled trial (RCT) published in the literature on this field. However, the published RCT was an open label study with no sham-controlled arm which could contribute to reporting bias and the treatment intensity might not be adequate. In our proposed study, we make a hypothesis that LiESWT and very early PDE5i can improve erectile function in patients after nerve-sparing radical prostatectomy.

DETAILED DESCRIPTION:
Urinary incontinence and erectile dysfunction (ED) are two most common complications after RP. Despite the advancement of prostate cancer treatment, erectile dysfunction post-prostatectomy remains as a significant morbidity especially for patients who are sexually active pre-operatively. PDE5i such as Tadalafil, Sildenafil remains the main form of penile rehabilitation with limited success. Non-invasive treatment such as Li-ESWT has proven to be a good treatment option mainly for vasculogenic ED. This study aims to investigate the effect of Li-ESWT treatment on post-prostatectomy ED, along with regular PDE5i.

Our hypothesis is that Low intensity extracorporeal shockwave therapy and very early PDE5i can improve erectile function in patients after nerve-sparing post-radical prostatectomy.

Eligible patients will be randomized to intervention arm (LiESWT treatment for 6 weeks + Tadalafil 5mg daily for 12 months) or controlled arm (sham therapy for 6 weeks + Tadalafil 5mg daily for 12 months). The device used in this study is Dornier Aries 2, with treatment protocol as described. The vacuum pump is an option for penile rehabilitation protocol at our institution due to its expensive cost. Penile vacuum pumps are allowed for voluntary use by all participants in both groups. A sub-group analysis will be conducted at the conclusion of the study.

Sexual outcomes will be assessed using IIEF (International Index of Erectile Function), EHS (Erectile Hardness Score) and Erectile Dysfunction Inventory of Treatment Satisfaction Score (EDITS) questionnaires at 1,3,6 and 12 months after completion of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent radical prostatectomy (open, laparoscopic or robotic-assisted) with nerve-sparing (unilateral or bilateral).
* Low / intermediate-risk prostate cancer
* PSA < 20 ng/ml
* Gleason score < 8
* Prostate cancer pathological stage </= T2b
* Sexually active with IIEF-5 score 3 18, with or without use of erectogenic aid / PDE5i.

Exclusion Criteria:

* Tumour upstaging beyond T2b
* Neurovascular bundle tissues bilaterally in the histopathological report.
* Scheduled treatment with pelvic radiotherapy and / or androgen deprivation therapy post-RP.
* Men with ED of neuropathological, endocrine or psychogenic origin.
* Previous pelvic surgery or radiation therapy.
* Patients with uncontrolled psychiatric conditions.
* Patients with major post-operative complications that could impact safety or effectiveness of ESWT.
* Patients with heart disease - unable to take PDE5i or prohibited from sexual activity.
* Patients on anticoagulation / antiplatelets except aspirin up to 100mg daily.
* Inflammation in the shockwave area or having penile pathology such as Peyronie's disease.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patient
Enrollment: 70 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Sexual Function | 12 months
  Measurement of average change in IIEF-5 score from baseline (pre-RP) to specified time-points at 1,3,6 and 12 months after completion of treatment - 22-25: No erectile dysfunction 17-21: Mild erectile dysfunction 12-16: Mild to moderate erectile dysfunction 8-11: Moderate erectile dysfunction 5-7: Severe erectile dysfunction 5 being the worst outcome

SECONDARY OUTCOMES:
Stretched Penile Length | 12 months
  Clinical measurement of change in stretched flaccid penile length from baseline specified time-points at 1,3,6 and 12 months after completion of treatment.
Urinary Function | 12 months
  Measurement of average change in EPIC questionnaire score from baseline (pre-RP) to specified time-points at 1,3,6 and 12 months after completion of treatment.
Safety and Adverse Events | 12 months
  Number of Participants With Treatment-Related Adverse Events as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Khor, ChM(Urol), Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Hospital Sultan Abdul Aziz Shah, Universiti Putra Malaysia (previously known as HPUPM), Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No